CLINICAL TRIAL: NCT06312514
Title: Status-neutral Community-based Multilevel Intervention to Address Intersectional Stigma and Discrimination, and Increase HIV Testing, PrEP, and ART Uptake Among YGBMSM in Ghanaian Slums: A Clustered Randomized Control Trial Protocol
Brief Title: Lafiya HIV-status Neutral Study - Protocol
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); University of Ghana (Other); Yale University (Other)
Responsible Party: Principal Investigator, Gamji Rabiu Abu-Ba'are, Assistant professor, University of Rochester
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00008615; R01NR021170 (NIH)
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: HIV Prevention and Care
Keywords: HIV testing; PrEP; ART; MSM; Ghana; HIV Status-Neutral; Slums; young men

STUDY DESIGN:
Intervention Model Description: intervention and waitlist control groups
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Participants will be young gay, bisexual and all other men who have sex men (YGBMSM) and providers from healthcare institutions working with (YGBMSM) who will receive the LAFIYA intervention.
  Interventions: Behavioral: LAFIYA
- Waitlist control group. (Experimental): Control arm for comparison who will receive the intervention after the intervention group
  Interventions: Behavioral: LAFIYA

INTERVENTIONS:
Behavioral: LAFIYA — The Lafiya intervention is a comprehensive program designed to address the intersectional stigma and discrimination challenges faced by marginalized communities, particularly among Gay, Bisexual, and other Men who have Sex with Men (GBMSM). It aims to enhance HIV prevention, care, and treatment outcomes, with a focus on increasing HIV self-testing (HIVST) uptake among these key populations in Ghanaian urban slum settings.

SUMMARY:
The primary objective of this study is to adapt and evaluate the feasibility of "Lafiya," which means "Wellness" in Hausa, a multilevel intersectional stigma & discrimination (ISD) and HIV testing intervention, to a status-neutral intervention to increase HIV testing, PrEP, and ART Uptake (HPART) among young gay, bisexual, and other men who have sex with men in Ghanaian slums. Specific objectives include, Assessing intersectional stigma and options for HPART implementation, Adapting Lafiya to a status-neutral intervention to address intersectional stigma and increase HPART uptake among YGBMSM, Test acceptance, feasibility, appropriateness, and preliminary efficacy of Lafiya to address intersectional stigma and increase HIVST uptake.

ELIGIBILITY:
Inclusion Criteria:

* YGBMSM FGD and IDI: To be eligible for FGD, the person must be between 18 to 25 years old, currently identify as a cis-gender man, have had sex with another man within 8 months before engaging with the recruitment team, and must reside within a slum community in the Accra metropolitan areas. To be eligible for IDIs, participants must self-disclose living with HIV.
* GBMSM civil society organizations FGD: The person must have experience providing GBMSM with HIV prevention and care services for at least one year. Must reside in the Accra metropolitan area.
* HCF staff FGDs: HCF staff are eligible to participate in the FGDs if employed at a study-participating facility.
* Anti-ISD Trained Nurses IDIs HCF staff are eligible to participate if they are trained in our previous interventions and have previously delivered them in a Ghanaian HCF.

Exclusion Criteria:

* YGBMSM FGD and IDI: Persons outside the age range of 18 to 25 years old, persons who do not identify as cis-gender men, persons who have not had sex with another man within 8 months before engaging with the recruitment team.
* GBMSM civil society organizations FGD: persons who do not have experience providing GBMSM with HIV prevention and care services for at least one year. Persons who do not reside within a slum community in the Accra metropolitan area (residence outside this area would be excluded).
* HCF staff FGDs: HCF staff are not eligible to participate in the FGDs if they are not employed at a study-participating facility.
* Anti-ISD Trained Nurses IDIs: HCF staff are not eligible to participate if they are not trained in our previous interventions and have not previously delivered them in a Ghanaian HCF.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 880 (Estimated)
Dates: Start 2025-04-20 (Estimated); Primary Completion 2028-08-29 (Estimated); Study Completion 2028-08-29 (Estimated)

PRIMARY OUTCOMES:
Change in HIV testing. | Baseline to 9 months
  We are going to collect the total number of HIV tests performed by all participants and report the mean change in numbers.
Change in PrEP Adherence. | Baseline to 9 months
  We will collect the total number of PrEP uptake and report the mean change in adherence ( mean change in urine tenofovir levels).
Change in ART Adherence | Baseline to 9 months
  We will assess changes in ART adherence among participants receiving HIV treatment, reporting mean changes in ART adherence (measured by HIV RNA levels).
Change in Treatment Self-Efficacy. | Baseline to 9 months
  We will assess changes in treatment self-efficacy among participants receiving HIV treatment, reporting mean changes in treatment self-efficacy scores. The scale will inquire into the experiences of treatment-related behaviors related to adhering to treatment plans, with responses categorized as "yes" or "no." The survey results are then analyzed by calculating the percentage change of participants who responded affirmatively (yes) to each question. The average percentage across all questions is calculated for an overall percentage.

SECONDARY OUTCOMES:
Percentage change in HIV stigmatizing attitudes. | Baseline to 9 months
  Using the HIV stigmatizing scale, participants will be provided with an 18-question survey that measures mean changes in HIV stigmatizing attitudes before and after the intervention.Each question will inquire into experiences of stigmatizing attitudes from others, with responses categorized as "yes" or "no." The survey results are then analyzed by calculating the percentage change of participants who responded affirmatively (yes) to each question. The average percentage across all questions is calculated for an overall percent.
Percentage change in reported sexual behavior stigma. | Baseline to 9 months
  Using the sexual behavior stigma scale, participants will be provided with a 13-question survey that measures the mean changes in perceived, anticipated, and enacted sexual behavior stigma.Each question inquires whether they agree or disagree with perceived, anticipated, and enacted sexual behavior stigma, with responses categorized as "yes" or "no." The survey results are then analyzed by calculating the percentage change of participants who responded affirmatively (yes) to each question. The average percentage across all questions is calculated to arrive at an overall percent score.
Percentage change in gender nonconformity stigma | Baseline to 9 months
  Using the Gender Nonconformity Stigma Scale, participants will be presented with a 10-item survey designed to assess attitudes towards gender nonconformity. This survey will measure the mean changes in perceptions of feminine mannerisms and their associated stigma.Each question inquires into their experiences of stigma from being gender non-conforming, with responses categorized as "yes" or "no." The survey results are then analyzed by calculating the percentage change of participants who responded affirmatively (yes) to each question. The average percentage across all questions is calculated to arrive at an overall percent score.
Percentage change in PrEP-related stigma | Baseline to 9 months
  Using the Youth PrEP-related Stigma Scale, participants will be provided with a 14-item survey that measures the mean changes in perceptions of PrEP-related, including misconceptions, fears, and judgments surrounding its use. Each question inquires into their experiences of PrEP-related Stigma, with responses categorized as "yes" or "no." The survey results are then analyzed by calculating the percentage change of participants who responded affirmatively (yes) to each question. The average percentage across all questions is calculated to arrive at an overall percent score.
Neighborhood stigma | Baseline to 9 months
  Participants will be provided with a 15-question survey that inquires into the rate at which they experienced unfair treatment within their neighborhood. Each question will inquire into experiences of unfair treatment, with responses categorized as yes or no. The survey results are then analyzed by calculating the percentage change of participants who responded yes to receiving unfair treatment in their neighborhood. The average percentage across all questions is calculated for an overall percent score.
Mean change in the Basic Needs Satisfaction | Baseline to 9 months
  The Basic Needs Satisfaction scale is a 6-question scale that asks participants general questions about experiences of feeling free within their community while identifying as YGMSM. The outcome measure will analyze changes in average scores over time. The Basic Needs Satisfaction Scale is scored on a scale ranging from 1 to 10, where 1 represents the lowest possible level of basic needs satisfaction, and 10 represents the highest.
Percentage of participants that reported healthcare climate stigma. | Baseline to 9 months
  Participants will be provided with a 15-question survey that inquires into the rate at which they experienced unfair treatment within the healthcare setting. Each question will inquire into experiences of unfair treatment, with responses categorized on a Likert scale ranging from strongly agree to disagree strongly. The survey results are then analyzed by calculating the percentage change of participants who responded affirmatively to unfair treatment they experience. The average percentage across all questions is calculated for an overall percent score.
Percentage of participants that reported Brief Resilience | Baseline to 9 months
  The Brief Resilience Scale is a 6-question survey that inquires into the level of resilience of participants. The scale includes statements that assess individuals' ability to bounce back and adapt positively to challenges and setbacks. Each question inquires into their ability to bounce back or cope with challenges, with responses categorized as "yes" or "no." The survey results are then analyzed by calculating the percentage change of participants who responded affirmatively (yes) to each question. The average percentage across all questions is calculated to arrive at an overall percent score.
Changes in Healthcare facility Intersectional stigma and discrimination. | Baseline to 9 months
  Using the adapted LGBTQ and Healthcare facility HIV stigma scales from Promoting Reductions in Intersectional StigMa (PRISM), Participants will be provided with a 22-item survey that measures changes in stigmatizing attitudes by health workers related to HIV stigma and gender non-conforming stigma. Each question inquires into their experience of intersectional stigma and discrimination, with responses categorized as "yes" or "no." The survey results are then analyzed by calculating the percentage change of participants who responded affirmatively (yes) to each question. The average percentage across all questions is calculated to arrive at an overall percent score.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ghana, Accra, Ghana

IPD SHARING:
Plan to Share IPD: Undecided
It may not be shared because of the stigma and discrimination facing LGBTQ-plus persons and known providers for the population in Ghana.

REFERENCES:
- [Derived] Abu-Ba'are GR, Torpey K, Guure C, Nelson LE, Jeon S, McMahon J, Leblanc NM, Shamrock OW, Zigah EY, Apreku A, Dakpui HD, Agbemedu GRK, Boakye F, Adu P, Attisoe A, Adjaka G. Status-neutral community-based multilevel intervention to address intersectional stigma and discrimination, and increase HIV testing, PrEP, and ART uptake among YGBMSM in Ghanaian Slums: A clustered randomized control trial protocol. Res Sq [Preprint]. 2024 May 30:rs.3.rs-4486078. doi: 10.21203/rs.3.rs-4486078/v1. PMID 38854081